CLINICAL TRIAL: NCT04571346
Title: A Two Paramedian Vaginal Incisions Versus the Standard Longitudinal Incision of Trans-Obturator Tape Procedure for Management of Urinary Incontinence
Brief Title: Female Sling Procedure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, assistant lecturer of Urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU R51/2019
Record Dates: First submitted 2020-09-19; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Urinary Incontinence,Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Female patients complaining of stress urinary incontinence will be selected for our study, at the urology department, Ain-shams University hospitals. Those patients will be randomized into 2 equal groups with a 1:1 ratio using sealed envelopes that will be prepared by the department's ethical committee, group 1 represents the classical TOT procedure while group 2 represents the 2 paramedian vertical incisions technique. Patients will be blinded to the type of intervention. Informed consent will be obtained for all patients before the surgery, Careful evaluation will be done including history taking, examination with a stress test and urodynamic study. Patients with neurological disease, pelvic organ prolapse, previous urethral or pelvic floor surgery will be excluded from our study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be blinded to the type of intervention as well as the data collector and the statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the classical TOT procedure (Active Comparator): performing the trans-obturator procedure through the standard vertical incision
  Interventions: Procedure: trans-obturator procedure
- 2 paramedian vertical incisions (Experimental): performing the trans-obturator procedure through a new technique of 2 paramedian vertical incisions
  Interventions: Procedure: trans-obturator procedure

INTERVENTIONS:
Procedure: trans-obturator procedure — TOT procedure will be done using silicon-coated polypropylene tape that will be inserted at the mid-urethral portion. In group 1, a classical vertical vaginal incision will be done proximal to the external urethral meatus with dissection along the axis of the urethra till the mid-urethral zone that is identified by palpating the urethral catheter balloon through the vaginal at the bladder neck, while in group 2, two paramedian incisions will be done 1cm long in the anterior vaginal wall 2 cm apart parallel to the urethra till identification of the mid-urethral portion, communication will be done between the two incisions 1 cm wide in this area creating a tunnel where the tape will be placed, this technique provides healthy tissues proximal and distal to the tape that allows more stabilization and less migration. The rest of the procedure is the same as the standard procedure of Trans-obturator outside-in tension-free technique.

SUMMARY:
In trans-obturator tape (TOT), tension and location of the tape in mid urethral zone are directly related to the postoperative clinical outcome. Recurrence of symptoms of stress urinary incontinence has been related to tape migration in previous studies. The study aimed to increase the success rate of TOT procedure through a new surgical technique using a 2 paramedian vaginal incisions.

DETAILED DESCRIPTION:
the investigator innovated a new technique that involves a 2 paramedian vaginal incisions that allow more tape stabilization with sparing the dissection along the whole urethra ensuring intact overlying tissues and to create a tunnel in between the 2 incisions to pass the tape, making it supported proximally and distally with normal undissected tissues.

the study aims to assess the success rate of TOT and tape migration using a new surgical technique versus the standard procedure using vertical incision.

ELIGIBILITY:
Inclusion Criteria:

* adult female patient complaining of pure stress incontinence confirmed by stress test of urodynamic study

Exclusion Criteria:

* Patients with neurological disease, pelvic organ prolapse, previous urethral or pelvic floor surgery will be excluded from our study.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — we evaluation the procedure of trans-obturator tape in female stress incontinence
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
tape migration | to be evaluated at 3rd month postoperative
  to evaluate TOT migration postoperative from the middle third of the urethra by trans-labial ultrasound
tape migration | to be evaluated at 6th month postoperative
  to evaluate TOT migration postoperative from the middle third of the urethra by trans-labial ultrasound
tape migration | to be evaluated at12th month postoperative
  to evaluate TOT migration postoperative from the middle third of the urethra by trans-labial ultrasound

SECONDARY OUTCOMES:
continence after surgery | to be evaluated at 3,6 and 12 month postoperative
  to evaluate success rate in treatment of stress urinary incontinence using stress cough test and urodynamic study
de-novo urgency | to be evaluated at 12 month postoperative
  appearance of urgency incontinence from patient symptomology evaluation whether present or not
vaginal erosion | to be evaluated up to 1 year post operative
  postoperative complication of TOT where vagina erosion may occur, (yes/no)
urine retention | to be evaluated in the first 24 hours postoperative
  postoperative complication of TOT ( present or not)

IPD SHARING:
Plan to Share IPD: No